CLINICAL TRIAL: NCT00834210
Title: Dapsone Gel 5% and Tazarotene Cream 0.1% Versus Tazarotene Cream 0.1% Monotherapy for Facial Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-ACZ0802
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Dapsone; tazarotene

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Active Comparator): Dapsone Gel 5% and Tazarotene Cream 0.1%
  Interventions: Drug: Dapsone
- 2 (Active Comparator): Tazarotene Cream 0.1%
  Interventions: Drug: Tazarotene

INTERVENTIONS:
Drug: Dapsone — Dapsone topical gel 5%, 1 pea-size amount BID x 12 weeks and Tazarotene Cream 0.1%, 1 pea-size amount QD x 12 weeks
  Other Names: Aczone Gel 5%; Tazorac Cream 0.1%
  Arms: 1
Drug: Tazarotene — Tazarotene Cream 0.1%, 1 pea-size amount QD x 12 weeks
  Other Names: Tazorac Cream 0.1%
  Arms: 2

SUMMARY:
A 12-week evaluation of the safety and efficacy of dapsone gel 5% when used with tazarotene cream 0.1% compared with tazarotene cream 0.1% monotherapy in treating moderate to severe facial acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Facial acne vulgaris characterized by the following: 30-100 facial inflammatory lesions; and 25-100 facial non-inflammatory lesions; stable disease, non-rapidly regressing facial acne vulgaris; and, 3 or more nodules and/or cysts (diameter of 1cm or greater). Female subjects of childbearing potential must have a negative pregnancy test at baseline and practice reliable method of contraception throughout the study

Exclusion Criteria:

* Non-compliance with washout period; history of clinically significant anemia or hemolysis; skin disease/disorder that might interfere with diagnosis or evaluation of acne vulgaris; allergy or sensitivity to any component of the test medications

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Fremont, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapsone Gel 5% and Tazarotene Cream 0.1%: Dapsone Gel 5% and Tazarotene Cream 0.1%
- Tazarotene Cream 0.1%: Tazarotene Cream 0.1%
Period: Overall Study
Arm/Group | Dapsone Gel 5% and Tazarotene Cream 0.1% | Tazarotene Cream 0.1%
Started | 86 | 85
Completed | 83 | 77
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapsone Gel 5% and Tazarotene Cream 0.1% | Tazarotene Cream 0.1% | Total
Number analyzed (Participants) | 86 | 85 | 171
Age Continuous [Median (Full Range); unit: years] | 17.8 [12.2 to 45.7] | 16.7 [12.1 to 42.9] | 17.2 [12.1 to 45.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 36 | 84
  Male | 38 | 49 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Inflammatory Lesion Counts (Papules,Pustules, and Nodules) at Week 12
Description: Change from baseline in inflammatory lesion count (papules, pustules and nodules) at week 12. Papules and nodules are round, solid elevations of the skin with no visible fluid; papules are smaller (less than 5 or 10 millimeters in width and depth) and nodules are larger (greater than 5 or 10 millimeters in width and depth). Pustules are small elevations of the skin containing cloudy material. A negative number change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT), which included all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Number of Lesions
Arm/Group | Dapsone Gel 5% and Tazarotene Cream 0.1% | Tazarotene Cream 0.1%
Number analyzed (Participants) | 86 | 85
Number of Lesions
  Baseline | 38.94 (11.67) | 40.78 (12.85)
  Week 12 | -25.77 (11.23) | -24.82 (14.06)

2. Secondary Outcome: Change From Baseline in Investigator Global Assessment at Week 12
Description: Change from baseline in the Investigator Global Assessment (IGA) at week 12. The IGA is a 5-point scale used by the investigator to assess overall acne severity, where 0 equals clear skin (no evidence of acne) and 4 equals severe acne. A negative number change from baseline indicates a reduction in acne severity (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT), which included all patients who started the study (randomized)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dapsone Gel 5% and Tazarotene Cream 0.1% | Tazarotene Cream 0.1%
Number analyzed (Participants) | 86 | 85
Scores on a scale
  Baseline | 2.93 (0.37) | 3.04 (0.36)
  Week 12 | -1.07 (0.96) | -0.96 (0.73)

3. Secondary Outcome: Change From Baseline in Overall Disease Severity at Week 12
Description: Change from baseline in overall disease severity at week 12. The overall disease severity was evaluated by the investigator using a 7-point scale to rate the overall acne severity (lesions, inflammation, facial redness and skin condition), where 0=no acne lesions and 6=most severe acne. A negative number change from baseline indicates a reduction in overall acne disease severity (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT), which included all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dapsone Gel 5% and Tazarotene Cream 0.1% | Tazarotene Cream 0.1%
Number analyzed (Participants) | 86 | 85
Scores on a scale
  Baseline | 4.03 (0.73) | 4.08 (0.69)
  Week 12 | -1.93 (1.11) | -1.63 (1.08)

4. Secondary Outcome: Change From Baseline in Non-Inflammatory Lesion Counts (Open and Closed Comedones) at Week 12
Description: Change from baseline in non-inflammatory lesion counts(open/closed comedones) at week 12. Comedones are small bumps on the skin (lesions) caused by acne and found at the opening of a skin pore. Open comedones (also known as blackheads) have a microscopic opening to the skin surface, while closed comedones (also known as whiteheads or "pimples") lack the opening to the skin. A negative number change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT), which included all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Number of lesions
Arm/Group | Dapsone Gel 5% and Tazarotene Cream 0.1% | Tazarotene Cream 0.1%
Number analyzed (Participants) | 86 | 85
Number of lesions
  Baseline | 46.42 (17.40) | 46.48 (16.86)
  Week 12 | -26.73 (15.08) | -21.74 (18.15)

ADVERSE EVENTS:
Arm/Group | Dapsone Gel 5% and Tazarotene Cream 0.1% | Tazarotene Cream 0.1%
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/85
Other Adverse Events (participants affected / at risk) | 8/86 | 5/85
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapsone Gel 5% and Tazarotene Cream 0.1% (N=86) | Tazarotene Cream 0.1% (N=85)
Cold (Infections and infestations) | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo